CLINICAL TRIAL: NCT06724458
Title: Skeletal Muscle Endurance Responses to Various Relative Loads of Dynamic Resistance Exercise with and Without Peripheral Blood Flow Occlusion
Brief Title: Resistance Exercise Blood Flow Restriction
Acronym: BFRCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Cameron Mitchell, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: BFRCL
Record Dates: First submitted 2023-06-09; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2023-06

CONDITIONS: Skeletal Muscle Endurance
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (12):
- 80% knee extension/80% barbell curl 1RM (Experimental): The load will be set to 80% of 1RM for the knee extension and 80% 1RM for the barbell curl
  Interventions: Other: Resistance exercise
- 40% knee extension/70% barbell curl 1RM (Experimental): The load will be set to 40% of 1RM for the knee extension and 70% 1RM for the barbell curl
  Interventions: Other: Resistance exercise
- 30% knee extension/60% barbell curl 1RM (Experimental): The load will be set to 30% of 1RM for the knee extension and 60% 1RM for the barbell curl
  Interventions: Other: Resistance exercise
- 25% knee extension/55% barbell curl 1RM (Experimental): The load will be set to 25% of 1RM for the knee extension and 55% 1RM for the barbell curl
  Interventions: Other: Resistance exercise
- 20% knee extension/50% barbell curl 1RM (Experimental): The load will be set to 25% of 1RM for the knee extension and 50% 1RM for the barbell curl
  Interventions: Other: Resistance exercise
- 15% knee extension/45% barbell curl 1RM (Experimental): The load will be set to 15% of 1RM for the knee extension and 45% 1RM for the barbell curl
  Interventions: Other: Resistance exercise
- 80% knee extension/80% barbell curl 1RM both with blood flow occlusion (Experimental): The load will be set to 80% of 1RM for the knee extension and 80% 1RM for the barbell curl with both being under peripheral blood flow occlusion
  Interventions: Other: Resistance exercise
- 40% knee extension/60% barbell curl 1RM both with blood flow occlusion (Experimental): The load will be set to 40% of 1RM for the knee extension and 60% 1RM for the barbell curl with both being under peripheral blood flow occlusion
  Interventions: Other: Resistance exercise
- 30% knee extension/60% barbell curl 1RM both with blood flow occlusion (Experimental): The load will be set to 30% of 1RM for the knee extension and 60% 1RM for the barbell curl with both being under peripheral blood flow occlusion
  Interventions: Other: Resistance exercise
- 25% knee extension/55% barbell curl 1RM both with blood flow occlusion (Experimental): The load will be set to 25% of 1RM for the knee extension and 55% 1RM for the barbell curl with both being under peripheral blood flow occlusion
  Interventions: Other: Resistance exercise
- 20% knee extension/50% barbell curl 1RM both with blood flow occlusion (Experimental): The load will be set to 20% of 1RM for the knee extension and 50% 1RM for the barbell curl with both being under peripheral blood flow occlusion
  Interventions: Other: Resistance exercise
- 15% knee extension/45% barbell curl 1RM both with blood flow occlusion (Experimental): The load will be set to 15% of 1RM for the knee extension and 45% 1RM for the barbell curl with both being under peripheral blood flow occlusion
  Interventions: Other: Resistance exercise

INTERVENTIONS:
Other: Resistance exercise — All arms will involve participants performing resistance exercise bouts of the described exercises. at the given loads, and with the stated flow condition

SUMMARY:
The number of repetitions able to be performed during resistance exercise is impacted by the load an individual is working against. Heavier loads lead to less repetitions being performed and lighter loads lead to more repetitions being performed. As the load gets progressively lighter, it is hypothesized that oxygen availability becomes an important factor for performance of maximum repetitions. Peripheral blood flow occlusion using exercise specific blood flow occlusion cuffs can allow for oxygen availability to be controlled by altering the amount of blood able to get to working muscles. To date, no study has examined the effect of varying exercise loads, from heavy to light, on maximum repetitions able to be performed with and without blood flow occlusion.

DETAILED DESCRIPTION:
The study aims to assess the difference in maximum repetitions performed at varying percentages of participants maximum strength and the impact peripheral blood flow occlusion has on performance

The study will take three weeks to complete with a total of six visits. The entire time commitment will be seven hours. During week 1 participants will visit the lab twice to perform baseline assessments of strength, endurance, muscle size and will also receive a resting thighs muscle biopsy. During weeks 2 and 3 participants will visit the lab twice per week to complete three out of twelve randomized exercise interventions per visit. The interventions are maximum repetitions at 80/40/30/25/20/15% of knee-extension one-repetition maximum as well as 90/70/60/55/50/45% of barbell curl one-repetition maximum; all of the listed conditions will be tested in a free-flow and blood flow occluded state (i.e., 12 total exercise interventions for the knee extension and 12 total exercise interventions for the barbell curl).

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and communicate in English
2. 19-30 years of age
3. All "No" answers on the Canadian Society for Exercise Physiology Get Active questionnaire or doctors' approval to participate
4. Untrained participants: no structured resistance and/or endurance training over the past 12-months (i.e., >2 hours per week of structured/periodized training)
5. Resistance trained participants: structured resistance training over the past 12-months (i.e., >2 hours per week of structured/periodized resistance training)
6. Endurance trained participants: structured resistance training over the past 12-months (i.e., >2 hours per week of structured/periodized endurance training)

Exclusion Criteria:

1. BMI lower than 18 or greater than 30
2. Current use of cigarettes or other nicotine devices
3. Any major uncontrolled cardiovascular, muscular, metabolic, and/or neurological disorders
4. Any medical condition impacting the ability to participate in maximal exercise
5. Type one or type two diabetes
6. Diagnosis of cancer or undergoing cancer treatment in the past 12 months
7. Taking blood-thinning medication or the presence of a bleeding disorder
8. Drug therapy with any drugs that alter skeletal muscle metabolism (i.e., Metformin, Benzodiazepines)
9. Lowest calculated exercise testing load is less than the lightest weight able to be provided by the lab gymnasium equipment (i.e., 36 pounds for the knee extension, and/or 33 pounds for the barbell curl)

Ages: 19 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2023-01-28 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Maximum knee extension repetitions | From weeks two to three in the study
  total repetitions completed for each load condition

SECONDARY OUTCOMES:
Maximum barbell curl repetitions | From weeks two to three in the study
  total repetitions completed for each load condition
Change in vastus lateralis oxygen saturation | From weeks two to three in the study
  The change in vastus lateralis oxygen saturation across each load condition
Correlation of muscle fiber size/type/distribution to maximum knee extension repetitions at 20% 1RM | From weeks two to three in the study
Correlation of mitochondrial content to maximum knee extension repetitions at 20% 1RM | From weeks two to three in the study
Correlation of capillary density to maximum knee extension repetitions at 20% 1RM | From weeks two to three in the study
Comparison of muscle fiber size/type/distribution, mitochondrial function, mitochondrial density, capillary density, absolute muscle size ,and VO2 max between participants of different training statuses | Week 3
Correlation of absolute muscle size to maximum knee extension repetitions at 20% 1RM/barbell curl repetitions at 45% 1RM | Weeks 1, 2, and 3
Correlation of absolute muscle size to maximum knee extension repetitions at 20% 1RM/barbell curl repetitions at 45% 1RM | Week 1
Correlation of absolute muscle size to maximum knee extension repetitions at 20% 1RM/barbell curl repetitions at 45% 1RM | Week 2
Comparison of absolute muscle size between sexes | Week 3
Comparison of capillary density between sexes | Week 3
Comparison of mitochondrial density between sexes | Week 3
Comparison of muscle fiber distribution between sexes | Week 3
Comparison of muscle fiber size between sexes | Week 3
Comparison of muscle fiber type between sexes | Week 3
Comparison of mitochondrial function between sexes | Week 3
Comparison of VO2 max between sexes | Week 3
Correlation of VO2 max to maximum knee extension repetitions at 20% 1RM | Week 1
Correlation of VO2 max to maximum knee extension repetitions at 20% 1RM | Week 2
Correlation of VO2 max to maximum knee extension repetitions at 20% 1RM | Week 3

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Gunn Pavilion, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
A plan has not yet been made to make individual participant data available to other researchers